CLINICAL TRIAL: NCT00650754
Title: A Randomized Double Blinded Trail of DHEA Supplementation for Treatment of Couples With Normal Hysterosalpingogram and Normal Semen Analysis and Evidence of Premature Ovarian Aging (POA).
Brief Title: Study of Oral Dehydroepiandrosterone(DHEA) to Treat Previously Unexplained Infertility
Acronym: DHEAFert
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Failure to recruit designed nuimebrt of subjects
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHR2008 1.0
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Primary Ovarian Insufficiency; Unexplained Infertility
Keywords: DHEA; Pregnancy
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHEA (Experimental): Dehydroepiandrosterone (DHEA) administered at a dose of 25 mg tid po. DHEA is a weak androgen produced naturally by the adrenal in men and women. DHEA production is diminished with increasing age. Peak levels of DHEA occur in the late teenage years.
  Interventions: Dietary Supplement: Dehydroepiandrosterone
- Placebo (Placebo Comparator): Blinded placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone — 25 mg PO TID
  Other Names: DHEA
  Arms: DHEA
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The experimental focus of this project is on the interaction of DHEA treatment on pregnancy in women with otherwise unexplained infertility and evidence of premature ovarian aging (POA).

DETAILED DESCRIPTION:
Recruitment:

Eligible patients will be recruited by advertising on the web and in newspaper. We will screen women under 38 years old with regular menstrual cycles and more than one year of infertility.

Experimental plan:

1. Informed consent
2. Baseline studies

   * Antral follicle counts on Day 2 - 3 of cycle
   * Day 3 Serum FSH, LH, E2, Prog, DHEA, DHEAS, testosterone, AMH, Fragile X
3. Randomization for pretreatment

   * Group A: DHEA (25 mg three times per day)
   * Group B: Placebo
4. Monitoring during treatment

   * All participants will have:
   * USG for follicle measurement
   * Repeat serum, FSH, E2, DHEA, DHEAS, testosterone, AMH monthly during treatment.
   * Physical examination
   * Completion of study questionnaire regarding possible androgen effects of treatment
5. Analysis plan:

   * Primary Outcome
   * Pregnancy
   * Pregnancy rates will be compared using logistic regression with age and pre-treatment AMH as covariates.
   * Secondary Outcomes
   * Endocrine Factors
   * Androgen side effects
   * Primary analysis. We will perform a factorial ANOVA for the two pretreatment factors DHEA and Placebo. Baseline AMH and age as main covariates
   * Secondary analysis.
   * Examine rate of change of estradiol and other endocrine response over the four cycles of pretreatment
   * Compare antral follicle counts across pretreatment cycles between groups
   * Compare possible androgen related effects
   * Power considerations:
   * Power assumptions: alpha 0.05; 80% power
   * Pregnancy rate for unexplained infertility is 2% per cycle.
   * Intervention will improve pregnancy rate to 5% per cycle.
   * Patients will be treated for 8 cycles.
   * Cumulative pregnancy rate for control patients - 13%
   * Cumulative pregnancy rate for Treated patients - 30%
   * Require 91 patients to complete treatment in each group.
   * Allow for 20% dropout ( 91* 1.2) will need 109 patients randomized to each group.
   * Randomization:

Randomization will be by permuted blocks in order to maintain an even distribution among the groups (because of the small numbers of participants)

* Human subjects issues
* Potential risks associated with DHEA use
* Potential risk of delay of treatment for 8 months and possible natural continued loss of fertility
* Informed consent issues

ELIGIBILITY:
Inclusion Criteria:

* >= 1 year of infertility
* < 38 years old
* Normal HSG
* Normal Semen analysis (Count >= 20 million/ motility > 50%/ Kruger morph > 14%.
* Regular menses
* Willingness to sign informed consent for study randomization
* Willingness to participate in 8 months of non-IVF will he him treatment.

Exclusion Criteria:

* Abnormal semen analysis
* Abnormal HSG
* Baseline FSH/E2 within normal age specific criteria
* Medical condition that would contraindicate pregnancy, ovulation induction or general anesthesia
* Family history of significant genetic disease, or factor V leiden thrombophilia
* Inability to present for monitoring visits
* Inability to follow medication instruction
* Desire to undergo other fertility treatments before completing eight months of this trial

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Live Birth | 24 months

SECONDARY OUTCOMES:
Endocrine effects | 12 months
Androgen side effects | 12 months
Clinical Pregnancy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Barad, MD, MS, Principal Investigator — Center for Human Reproduction; Norbert Gleicher, MD, Study Chair — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

REFERENCES:
- See also: Center for Human Reproduction — http://www.centerforhumanreprod.com/